CLINICAL TRIAL: NCT02283905
Title: Case Series of Continuously-infused Amphotericin-B and Follow-up Voriconazole Therapy for Severe Blastomycosis Pulmonary Infections
Brief Title: Amphotericin-B and Voriconazole for Pulmonary Blastomycosis
Acronym: BLASTO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment numbers of patients
Sponsor: University of Manitoba (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Robert Ariano, Professor of Pharmacy and Medicine, Critical Care Pharmacist, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2014:032
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Blastomycosis
Keywords: amphotericin-B; continuously infused; voriconazole
MeSH Terms: conditions — Blastomycosis | interventions — Amphotericin B; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amphotericin-B and Voriconazole (Other): Treatment with a 24 hour continuous infusion of amphotericin B deoxycholate at 1.0 mg/kg/day for a total dose of at least 1 g (i.e. ~ 14 days); and then the patient is stepped down to voriconazole 6 mg/kg i.v. q12h for 2 doses, then 4 mg/kg q12h either i.v. or orally as appropriate. The oral dose will be rounded for convenience to either the 200 mg or 400 mg tablet twice daily.
  Interventions: Drug: amphotericin-B; Drug: voriconazole

INTERVENTIONS:
Drug: amphotericin-B — continuously infused
  Other Names: Fungizone
Drug: voriconazole — intravenously or orally administered
  Other Names: Vfend

SUMMARY:
All patients with pulmonary blastomycosis requiring mechanical ventilation will have their blood concentrations measured for the antifungal drugs, amphotericin-B and voriconazole; as well as an analysis of the susceptibility of their infecting species of blastomyces. This information will then be analyzed relative to their rate of clinical recovery from this serious fungal infection.

DETAILED DESCRIPTION:
To evaluate six intensively studied patients admitted to medical intensive care with pulmonary blastomycosis requiring mechanical ventilation. Interventionally, all patients will receive continuously infused amphotericin-B (1 mg/kg/d); and then stepped down to oral or i.v. voriconazole once clinically responding. Blood will be sampled for amphotericin-B concentrations for the 3 first days (i.e. one blood sample per day); and when eventually changed over to voriconazole (i.e. generally after a total dose of 1 g has been reached of Amphotericin-B; as per usual practice). Once switched to oral or intravenous voriconazole, at the treating physicians discretion, then blood would once again be sampled for the next 3 days for voriconazole concentrations. MIC's of the infecting blastomyces would also be analyzed. The fungal isolate would be sent off to the Fungus Testing Laboratory at the University of Texas in San Antonio for susceptibility testing.

Clinical response to therapy relative to their initial pharmacokinetic and pharmacodynamic indices for amphotericin-B (i.e. daily free maximal concentration divided by the MIC) would be assessed in these 6 intensively studied patients. Clinical parameters assessed would be 1). time to fever defervescence; 2). time to white cell count resolution, and 3). improvements in respiratory gas exchange (i.e. specifically the rate of rise of the pressure of arterial oxygen (Pa02) divided by the fraction of inspired oxygen (Fi02) delivered through the ventilator (or PF ratio).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients 18 years of age or older admitted to the intensive care units of St. Boniface General Hospital with a diagnosis of acute pulmonary blastomycosis requiring mechanical ventilation.

Exclusion Criteria:

* The patient's data will be excluded if they die within 3 days of hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
The concentration-time profile of antifungals during treatment relative to the level of susceptibility of the infecting organism | within the first month of therapy

SECONDARY OUTCOMES:
Clinical recovery - as assessed by time to fever defervescence; and white blood cell (WBC) count resolution | 2 to 3 days
  Temperature would be assessed at least 4 times daily; and once there was a sustained temp < 38 degrees Celsius the timing would stop. WBC would be assessed at least twice daily and once the count fell less than 12,000 the timing would stop.
Clinical recovery - time to discontinuation of mechanical ventilation | less than 7 days
  Defined as the interval between initiation of amphotericin-B infusion and when the patient was considered ready for extubation. A patient was considered ready for extubation if awake or arousable, neurologically intact, cooperative and comfortable, fraction of inspired oxygen (FiO2) < or = 0.4, positive end-expiratory pressure (PEEP) < or = 5 cm water (H2O); and at the attending physicians discretion. Patient status will be assessed for extubation at least once daily.
Clinical recovery - time to respiratory dysfunction resolution | less than 4 days
  The daily assessment of the lowest pressure of arterial oxygen divided by the fraction of inspired oxygen (PF ratio = Pa02/Fi02) to detect the time until the PF ratio exceeds 200

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Ariano, Pharm.D., Principal Investigator — St. Boniface Hospital
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapman SW, Dismukes WE, Proia LA, Bradsher RW, Pappas PG, Threlkeld MG, Kauffman CA; Infectious Diseases Society of America. Clinical practice guidelines for the management of blastomycosis: 2008 update by the Infectious Diseases Society of America. Clin Infect Dis. 2008 Jun 15;46(12):1801-12. doi: 10.1086/588300. PMID 18462107
- [Background] Chowfin A, Tight R, Mitchell S. Recurrent blastomycosis of the central nervous system: case report and review. Clin Infect Dis. 2000 Jun;30(6):969-71. doi: 10.1086/313828. PMID 10880319
- [Background] Ariano RE, Mitchelmore BR, Lagace-Wiens PR, Zelenitsky SA. Successful treatment of pulmonary blastomycosis with continuously infused amphotericin B deoxycholate after failure with liposomal amphotericin B. Ann Pharmacother. 2013 Jun;47(6):e26. doi: 10.1345/aph.1R703. Epub 2013 May 14. PMID 23673538
- [Background] Eriksson U, Seifert B, Schaffner A. Comparison of effects of amphotericin B deoxycholate infused over 4 or 24 hours: randomised controlled trial. BMJ. 2001 Mar 10;322(7286):579-82. doi: 10.1136/bmj.322.7286.579. PMID 11238151